CLINICAL TRIAL: NCT07236034
Title: ARISe at UMass Chan: Remote Eye Tracking Study of Vaccine Messaging in Rural Populations
Brief Title: ARISe at UMass Chan
Acronym: ARISe
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Grace Ryan, Assistant Professor, University of Massachusetts, Worcester
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00002075; 1U48DP006883-01 (NIH)
Record Dates: First submitted 2025-10-01; First posted 2025-11-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Vaccination; Vaccination Promotion
Keywords: Message perceptions; Vaccination; Immunization

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of 14 conditions and view two messages within each.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Arm 1: Peer message, 7C Construct 1 (Experimental): This arm will include messages with a "peer" influence as the source and the construct of "confidence" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 2: Professional source, 7C Construct 1 (Experimental): This arm will include messages with a "professional" influencer as the source and the construct of "confidence" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 3: Peer message, 7C Construct 2 (Experimental): This arm will include messages with a "peer" influence as the source and the construct of "complacency" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 4: Professional message, 7C Construct 2 (Experimental): This arm will include messages with a "professional" influence as the source and the construct of "complacency" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 5: Peer message, 7C Construct 3 (Experimental): This arm will include messages with a "peer" influence as the source and the construct of "constraints" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 6: Professional message, 7C Construct 3 (Experimental): This arm will include messages with a "professional" influencer as the source and the construct of "constraints" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 7: Peer message, 7C Construct 4 (Experimental): This arm will include messages with a "peer" influencer as the source and the construct of "calculation" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 8: Professional message, 7C Construct 4 (Experimental): This arm will include messages with a "professional" influencer as the source and the construct of "calculation" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 9: Peer message, 7C Construct 5 (Experimental): This arm will include messages with a "peer" influencer as the source and the construct of "collective responsibility" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 10: Professional message, 7C Construct 5 (Experimental): This arm will include messages with a "professional" influencer as the source and the construct of "collective responsibility" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 11: Peer message; 7C Construct 6 (Experimental): This arm will include messages with a "peer" influencer as the source and the construct of "compliance" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 12: Professional message, 7C Construct 6 (Experimental): This arm will include messages with a "professional" influencer as the source and the construct of "compliance" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 13: Peer message, 7C Construct 7 (Experimental): This arm will include messages with a "peer" influencer as the source and the construct of "conspiracy" as the message.
  Interventions: Behavioral: Exposure to source and message content
- Arm 14: Professional message, 7C Construct 7 (Experimental): This arm will include messages with a "professional" influencer as the source and the construct of "conspiracy" as the message.
  Interventions: Behavioral: Exposure to source and message content

INTERVENTIONS:
Behavioral: Exposure to source and message content — Within each arm, participants will be exposed to two messages each of which are delivered by the same source (peer or professional) and have message content related to one of the 7C Constructs.

SUMMARY:
The goal is to identify the most impactful strategies for capturing attention and enhancing effectiveness of vaccine promotion messages. This will be done using an online survey that employs remote eye-tracking and self report measures to evaluate response to sample vaccine promotion social media content in rural populations in New England. Participants will be randomly assigned into one of 14 conditions in a 2(source: expert vs. influencer) by 7 (themes: constructs from 7C Vaccine Framework) experiment and view sample messages and then answer questions about their attitudes and beliefs while being monitored for eye-tracking.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+
* Living in New England state (CT, MA, ME, NH, VT RI) in a zip code as defined by each individual state's definition of rural
* Able to read and write in English
* Access to an internet connected computer or laptop with a web-camera

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Source credibility | Immediately after viewing each message
  Participants' perception of the credibility of the message source will be assessed using a 7-point Likert scale measured across four items. Participants will be asked to rate the following four items on this scale: To what extent do you believe the source of the message to be… (1=not at all, 7=very much so)
  1. Fair
  2. Accurate
  3. Telling the whole story
  4. Trustworthy
  Unit of measure: Scale score 1-7, mean
Perceived Message Effectiveness | Immediately after viewing each message
  Perceived message effectiveness will be measured using six items (worth remembering, grabs attention, powerful, informative, meaningful, convincing), each rated on a 7-point Likert scale. The outcome will be the mean of these six ratings for each participant, then averaged by experimental condition.
  To what extent is… (1=not at all, 7=very much so)
  1. The message worth remembering
  2. The message grabs attention
  3. This message powerful
  4. This message informative
  5. This message meaningful
  6. This message convincing Unit of Measure: Scale score (1-7, mean across items)
Visual attention | During message viewing ( immediately post-randomization, prior to completion of post-message survey)
  Visual attention, quantified as mean dwell time in milliseconds, will be measured using remote eye-tracking while participants view vaccine promotion messages. Dwell time will be calculated for pre-specified Areas of Interest (AOIs) during the message viewing period. Higher dwell times indicate greater visual attention to the AOIs.
  Unit of measure: mean dwell time in milliseconds per message
Message reactance | Immediately after viewing each message
  Reactance will be assessed using four items (irritated, angry, annoyed, aggravated), rated 0 ("None of this feeling") to 4 ("A great deal of this feeling"). The mean reactance score will be calculated for each participant.
  How much did this message make you feel the following way? Response options: 0 (None of this feeling) to 4 (A great deal of this feeling).
  1. Irritated
  2. Angry
  3. Annoyed
  4. Aggravated
  Unit of Measure: Scale score (0-4, mean across items)
Information sharing intentions | Immediately after viewing each message
  Description: Assessed with 6 items regarding interpersonal and online sharing, rated 1 (Strongly disagree) to 5 (Strongly agree). The mean score across items will be reported per participant and per condition.
  Rate with the following statements on a scale from 1 (Strongly disagree) to 5 (Strongly agree).
  Interpersonal setting
  1. I would be willing to share this information with others.
  2. I would talk with others about this message.
  3. I would point others in a direction where they could read this message.
     Online setting
  4. I would be willing to post a link to this information on my social media.
  5. I would like a social media post with this information.
  6. I would share a social media post with this information.
  Unit of Measure: Scale score (1-5, mean across items)

SECONDARY OUTCOMES:
Vaccine perceptions | Assessed at baseline (prior to message exposure) and immediately post-intervention (after message exposure)
  Vaccine perceptions will be measured using an 8-item scale, administered pre- and post-message exposure. Items are rated from 1 (Strongly disagree/very negative) to 7 (Strongly agree/very positive). Higher scores indicate more positive vaccine perceptions. The outcome will be the mean change in score from pre- to post-exposure.
  Unit of Measure: Scale score (1-7, mean change)

CONTACTS AND LOCATIONS:
Overall Officials: Grace W Ryan, PhD, MPH, Principal Investigator — University of Massachusetts Chan Medical School
Locations (1):
- University of Massachusetts Chan Medical School, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Per the data management plan, datasets and codebooks will be provided to individual researchers upon reasonable request.